CLINICAL TRIAL: NCT04247295
Title: RCT Comparing the Efficacy of POP Cast vs Woodcast for Distal Radial Fractures in Children.
Brief Title: Comparison of Woodcast vs Traditional Cast in Distal Radius Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCH-2187
Record Dates: First submitted 2020-01-03; First posted 2020-01-30 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Bone Fracture
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Intervention Model Description: 2 arms of randomised treatment methods, each participant will be either assigned to the traditional cast or the woodcast assigned.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wood cast (Experimental): Participants will be trialling the woodcast plaster method
  Interventions: Device: Woodcast
- Traditional Cast (Placebo Comparator): Traditional cast used to be compared to.
  Interventions: Device: Traditional Cast

INTERVENTIONS:
Device: Traditional Cast — Application of a traditional cast
  Arms: Traditional Cast
Device: Woodcast — Application of a woodcast
  Arms: Wood cast

SUMMARY:
The investigators project is a randomised controlled trial that will compare the efficacy of the traditional casting method against the woodcast splint in distal radial fracture. After the investigators have taken consent and the patients have agreed to be a part of the project, the investigators will randomly divide the participants into two groups. One with the traditional cast and one with the wood cast. The difference will be measured by using the EQ-5D-Y tool alongside the use of the DASH score and our own questionnaire.

The study will take place over the following year with the Sheffield Children's Hospital being the only site involved. Woodcast products have the CE declaration of conformity which is covered for the use in children, and apart from the type of cast the child is given, the course of treatment is the same for both group

DETAILED DESCRIPTION:
Distal radial fractures are a very common fracture. Without good plaster immobilisation these fractures are prone to slipping. As a result, patients may end up with surgical treatment which would otherwise not be needed if the plaster were to hold the fracture position adequately. If one was shown to be better compared to the other, then all hospitals could start to use a more effective treatment.

With traditional casting, some of the details of the fracture are missed due to the shadowing on the x-ray. The woodcast aims to reduce this shadowing, allowing a more detailed image of the fracture and hopefully a better outcome. Problems may arise with the plaster cast, at one or two week scans, in which the cast may need to be removed for imaging, this could lead to displacement of the fracture effecting the outcome. Woodcast would potentially not need to be removed or is easily removed due to the fact that it is not a complete cast and so would hopefully improve the outcomes for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 3 and 16 that present with a distal radial fracture.

Exclusion Criteria:

* Patients with underlying physical and learning disabilities.
* Patients with significant co-morbidities that would put the patient at risk of extra distress.
* Pathological fractures for instance Osteogenesis Imperfecta, metabolic bone diseases etc...
* Patients who aren't fluent in English as we only have questionnaires available in English.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2017-12-07 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Woodcast effectiveness measured by self designed patient response questionnaire. Score not reported on a scale | 3 months
  Whether the woodcast is comfortable to the patient
Woodcast effectiveness versus traditional cast | 3 months
  To measure the displacement of the fracture seen on the x-ray, comparing those in the traditional cast and those in the Woodcast.
Woodcast effectiveness | 3 months
  Whether the cast needs to be changed during the course of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Facility, Sheffield Childrens Hospital, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No